## The Elders' Resilience Curriculum NCT06045273 8/1/2023



## JOHNS HOPKINS BLOOMBERG SCHOOL OF PUBLIC HEALTH ASSENT FORM -AIM 3 SURVEY

Study Title: The Elders' Resilience Curriculum: Toward Building Empirical Evidence Around a Culturally-

Grounded, Strengths-Based Intervention

Principal Investigator: Dr. Victoria O'Keefe

**IRB No.:** 00018615

PI Version Date: 2 / 08.03.2023

Hello, I am [Data Collector Name] from Johns Hopkins Center for Indigenous Health and would like to talk to you about a research study we are doing. A research study is a way to learn about something. We want to learn about what you think when the Elders come teach in your classroom at school, and how the Elders teaching affects you. We would like you to join this study because you are between the ages of 9-14, in a school where the Elders' Resilience Curriculum program is being delivered, and you are participating in the Elders' Resilience Curriculum program.

If you want to join this study, you will fill out three surveys.

- You will fill out the surveys at school in your classroom. The first survey you fill out will be in the fall,
   then you will fill out a survey again in January, and the third survey in May. You will get a \$25 gift card
   for every survey that you fill out.
- The surveys will ask you questions about things like your health, how you feel connected to people and your culture, how much you speak Apache, and how you are doing at school.
- You may skip any questions in the survey that you do not want to answer.
- The survey questions do not ask you about negative things. If you do feel uncomfortable while filling out the survey, we will have people nearby who can help you.
- We will keep all of the answers you share in the survey private and will not share it with your parents, classmates, or teachers. All of the people who work on this study are trained to keep your information safe and private.
- We do not know if you will be helped by being in this study. We might learn something that will help other youth live strong healthy lives.

You do not have to join this study. It is up to you. You can say okay now, and you can change your mind later. All you have to do is tell us. No one will be mad at you if you change your mind.

1 450 1 01 4



| Do you have any questions? | |
|---|---|
| Would you like to join the study? | |
| If you want to join this study, please sign your name. We will give you a copy of this form to keep for yourself. | |
| Participant Name (print) | Date |
| | D.L. |
| Participant Signature | Date |
| Γο be completed by study staff: | |
| Name of staff obtaining assent (print) | <br>Date |
| J (1 / | |

Date

Signature of staff obtaining assent